CLINICAL TRIAL: NCT05761483
Title: Endoscopic Management of Non-anastomotic Biliary Strictures Following Liver Transplantation. Registry of the Italian Society of Digestive Endoscopy.
Brief Title: Endoscopic Management of Non-anastomotic Biliary Strictures Following Liver Transplantation.
Acronym: STEBINANSIED
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Tringali Andrea, MD, PhD, Assistant Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2766
Record Dates: First submitted 2023-02-25; First posted 2023-03-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant Disorder; Ischemic Cholangiopathy; Non-anastomotic Biliary Stricture; Biliary Stricture; Biliary Stents (Plastic)
Keywords: ERCP; Biliary stents; Liver transplantation; Ischemic cholangiopathy
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ERCP — Endoscopic Retrograde Cholangiopancreatography, placement of stents using a duodenoscope and making an access through the papilla of Vater
  Other Names: Biliary stents placement

SUMMARY:
The study will evaluate the results of endoscopic treatment of NON-anastomotic biliary strictures following liver transplantation

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Non anastomotic biliary strictures diagnosed by direct cholangiogram (T-tube) or MRCP
* Stricture involving the hepatic hilum until secondary branches
* Increase of liver function tests
* Signature of the informed consent

Exclusion Criteria:

* Previopus endoscopic or percutaneous treatments
* Patient candidate to metal stents placement
* Previous surgery resulting in altered anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that underwent liver transplantation and has a diagnosis of biliary strictures secondary to ischemic cholangiopaty (biliary stenoses involving bile ducts of the donor and extending to the hilum)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of endoscopic treatment of non-anastomosis biliary strictures | 2 Years follow-up
  Evaluate biliary stricture resolution rate

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tringali, MD, PhD, Principal Investigator — Fondazione Policlinico Gemelli IRCCS, Rome, Italy
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No